CLINICAL TRIAL: NCT07307092
Title: Comparison of Intramuscular Progesterone and Rectal Progesterone in the Prevention of Preterm Labour in Patients Undergoing Cervical Cerclage: A Randomized Controlled Trial
Brief Title: Intramuscular vs Rectal Progesterone in Preventing Preterm Labour After Cervical Cerclage
Acronym: PROCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hina Mukhtar (Other)
Responsible Party: Sponsor-Investigator, Hina Mukhtar, DR, Combined Military Hospital (CMH) institute of Medical Sciences Bahawalpur Pakistan
Organization: Combined Military Hospital (CMH) institute of Medical Sciences Bahawalpur Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMH-OBG-RCT-2025-01
Record Dates: First submitted 2025-12-13; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Preterm Labour; Cervical Insufficiency; Pregnancy, High-Risk
Keywords: Interventions; Population; Study design; Clinical focus
MeSH Terms: conditions — Obstetric Labor, Premature; Uterine Cervical Incompetence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intramuscular Progesterone Group (Experimental): Participants in this group received intramuscular progesterone (hydroxyprogesterone caproate) 250 mg once weekly, starting from 16 weeks until 36 weeks of gestation, following cervical cerclage. The injections were administered in the gluteal region under aseptic conditions. The purpose of this intervention was to maintain uterine quiescence and reduce the risk of preterm labour in high-risk pregnancies after cerclage.
  Interventions: Drug: Intramuscular Progesterone; Drug: Rectal Progesterone
- Rectal Progesterone Group (Experimental): Participants in this group received rectal progesterone suppositories 400 mg once daily, starting from 16 weeks until 36 weeks of gestation, following cervical cerclage. The suppositories were self-administered at bedtime. The aim of this intervention was to provide sustained progesterone support for maintaining uterine relaxation and reducing the risk of preterm labour after cerclage.
  Interventions: Drug: Intramuscular Progesterone; Drug: Rectal Progesterone

INTERVENTIONS:
Drug: Intramuscular Progesterone — Hydroxyprogesterone caproate 250 mg administered intramuscularly once weekly from 16 to 36 weeks of gestation following cervical cerclage. Used to maintain uterine quiescence and prevent preterm labour.
Drug: Rectal Progesterone — Micronized progesterone 400 mg suppository administered rectally once daily from 16 to 36 weeks of gestation following cervical cerclage. Intended to provide sustained progesterone support and prevent preterm labour.

SUMMARY:
Preterm labour is a major cause of neonatal morbidity and mortality worldwide. Progesterone supplementation is known to help reduce the risk of preterm birth in high-risk women. This randomized controlled trial compared the effectiveness of intramuscular progesterone and rectal progesterone in preventing preterm labour among pregnant women who had undergone cervical cerclage. The study aimed to determine which route of progesterone administration provides better pregnancy prolongation and improved neonatal outcomes.

DETAILED DESCRIPTION:
Background:

Preterm labour remains one of the leading causes of perinatal mortality and long-term neonatal complications. Cervical insufficiency, often managed by cervical cerclage, is a recognized risk factor for preterm birth. Progesterone supplementation helps maintain uterine quiescence and cervical integrity, but the optimal route of administration after cerclage is not well established.

Objective:

To compare the efficacy of intramuscular progesterone versus rectal progesterone in preventing preterm labour among women who underwent cervical cerclage.

Methods:

This single-centre, randomized controlled trial was conducted in the Department of Obstetrics & Gynecology, Bahawal Victoria Hospital, Bahawalpur, Pakistan. Eligible women with singleton pregnancies who had undergone cervical cerclage were randomly assigned to receive either weekly intramuscular progesterone (250 mg) or daily rectal progesterone suppositories (400 mg) from 16 to 36 weeks of gestation. The primary outcome was the incidence of preterm labour before 37 weeks. Secondary outcomes included gestational age at delivery, neonatal birth weight, NICU admission, and maternal side effects.

Significance:

This study provides evidence on the comparative effectiveness of two commonly used routes of progesterone administration in women with cerclage, aiming to identify the safer and more convenient regimen for prolonging pregnancy and improving neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

Pregnant women aged 18-45 years

Singleton pregnancy

Gestational age between 16 and 24 weeks at enrollment

Diagnosed with cervical insufficiency and scheduled for or recently undergone cervical cerclage

Willing to receive progesterone therapy and provide written informed consent

Exclusion Criteria:

Multiple pregnancy

Known fetal anomalies

Severe maternal comorbidities (e.g., hypertension, diabetes, cardiac disease)

History of allergy or hypersensitivity to progesterone or related compounds

Contraindications to progesterone use

Women who declined to participate or were non-compliant with follow-upInclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 820 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-04-25 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Frequency of Preterm Birth (<37 Weeks) | 16-36 weeks until delivery

SECONDARY OUTCOMES:
Gestational Age at Delivery | At delivery
Neonatal Birth Weight | At birth
Apgar Scores at 1 and 5 Minutes | Immediately post-delivery
NICU Admission Rate | Within 24 hours of birth
Maternal Adverse Effects | During treatment period (16-36 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Hina Mukhtar, MBBS, Principal Investigator — CMIS Bahawalpur
Locations (1):
- CIMS Bahawalpur, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No